CLINICAL TRIAL: NCT03735407
Title: Evaluation of Safety, Usability and Subject Compliance While Using Check- Cap's C-Scan System for Providing Structural Information on Colonic Polypoid Lesions and Masses
Brief Title: Safety,Usability and Compliance of Using C-Scan System for Providing Information on Colonic Polypoid Lesions and Masses
Acronym: C-Scan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-SY-02-0096
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, Multi-center, Single-arm, safety study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- C-Scan procedure (Experimental): Subjects who are at high or at average risk for developing CRC and who are scheduled for optical colonoscopy will undergo C-Scan procedure
  Interventions: Device: C-Scan procedure

INTERVENTIONS:
Device: C-Scan procedure — The subjects will be connected to the C-Scan Track and after successful system's activation. The subject will be asked to ingest the C-Scan Capsule with some water, contrast media The subject will be required to ingest daily dose (3 X 15 ml) of contrast media. Capsule procedure is completed upon capsule excretion.
  o Collecting procedure related data: Technical performance in normal daily routine, Segmental transit time,Procedure duration, Number of Bowel movements , Similarity between C-Scan results and colonoscopy Etc,
  Other Names: data collection to improve the product's algorithm

SUMMARY:
Protocol Title: Evaluation of safety, usability and subject compliance while using Check- Cap's C-Scan System for providing structural information on colonic polypoid lesions and masses Study Design: Prospective, Multi-center, Single-arm, safety study Purpose: To demonstrate the safety of the Check-Cap C-Scan System Study Centers: Up to two (2) centers located in the United States Number of Participants: 45 healthy subjects Investigational Device: Check-Cap's C-Scan System comprises C-Scan Capsule, C-Scan Track and C-Scan View.

Primary Objective: To evaluate the safety of the Check-Cap C-Scan System Secondary Objectives: a. To evaluate subject's compliance b. To evaluate subject's satisfaction c. To collect data to improve the product's algorithm

DETAILED DESCRIPTION:
Overall Design: Up to 45 healthy subjects will participate in this study. Subjects to be enrolled in this study are indicated and scheduled to undergo optical colonoscopy based on the following symptoms or by being classified as higher than average risk based on one or more of the following:

* Surveillance - Significant findings in previous optical colonoscopy
* Diagnostic - Polyps detected in virtual colonoscopy referred for polypectomy
* Diagnostic - Polyps detected in previous optical colonoscopy (community setting) referred for polypectomy
* Diagnostic - Positive FIT (Fecal Immunochemical Test)
* Diagnostic - one or more of the typical symptoms:
* abdominal pain
* Change in bowel habits
* Anemia or overt bleeding in stool
* Significant weight loss
* First degree relatives of CRC (Colo-Rectal Cancer)subjects Alternatively, average risk based on their age and demographics referred for screening for polyps

Each subject will receive a comprehensive explanation regarding the study nature. During this process, and per ethical committee approval, subjects may be asked several questions (over the phone) regarding their medical background for preliminary assessment of eligibility. Once informed consent is obtained, a thorough evaluation of subject's eligibility will be performed based on inclusion / exclusion criteria.

Eligible subjects will be required to undergo FIT procedure, per package insert instructions, within pre-defined timelines. All subjects will be scheduled to undergo capsule procedure, to be followed later on with optical colonoscopy procedure.

One to three days following end of C-Scan procedure the subjects will be contacted by phone by the clinical coordinator to follow-up on the subject well-being. Same follow-up procedures will be applied one to three days following Optical Colonoscopy procedure. Medical history and concomitant medication information will be collected for all subjects.

Study Duration: The duration of study participation for each subject is expected to be approximately 8-10 weeks. The total study duration across all patients is expected to be approximately 6 months, dependent upon subject recruitment rate.

C-Scan Procedure: Subjects will be instructed to skip breakfast or lunch on the day of C-Scan Capsule ingestion to expedite gastric passage. Liquids are allowed.

The subjects will be connected to the C-Scan Track and after successful system's activation (BIT - built in test), the subject will be asked to ingest the C-Scan Capsule with some water, contrast media (GE Omnipaque 350) and non-soluble fiber, in the presence of a physician investigator or designee. The subject will also be provided with an RF watch. A representative of the sponsor will attend the ingestion procedure, as needed to assure proper activation.

Post ingestion, the subject will receive detailed instructions about the daily routine and activities as well as use of the RF watch and then will be discharged home with written instructions on the procedure Instructions for use (IFU), daily diary, FIT kit and capsule return kit.

FIT Procedure: All subjects will be required to perform FIT procedure using [OC-Light] FIT Kit prior or during the capsule procedure Capsule Return: Capsule procedure is completed upon capsule excretion or system auditory indication of 'End of Procedure'. Subjects will be instructed to inform the study coordinator or designee upon capsule excretion

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at the age of 40-80 years' old.
2. Subject provided signed informed consent.
3. Subject is willing and able to comply with the specified study requirements and follow-up evaluations, and can be contacted by telephone.
4. Subjects able and agrees to undergo colonoscopy procedure.
5. BMI > 22 and ≤ 35.
6. Maximum body (abdominal) circumference < 120 cm.
7. Has at least 3 bowel movements per week
8. A colonoscopy procedure is pre-scheduled within 60 days

Exclusion Criteria:12.3 Exclusion Criteria

1. Known history of dysphagia or other swallowing disorders.
2. History of the followings: Inflammatory Bowel Disease (IBD) including Crohn's disease or Ulcerative, Colitis, Meckel's Diverticulum, Bowen Hernia, known fistulas or strictures (doctors' discretion), or a history of small bowel obstruction.
3. Known motility disorders:

i. Chronic Constipation: less than 3 bowel movements/week, w/out the use of laxatives.

ii. Delayed gastric emptying. iii. Narcotic use d. Prior history of abdominal surgery that might cause bowel strictures leading to capsule retention, as determined by physician discretion with the exception of appendectomy, cholecystectomy and hysterectomy e. Any condition believed to have an increased risk for capsule retention, strictures, bowel adhesion or other obstacles to free passage of the capsule (such as intestinal tumors, radiation enteritis) or incomplete colonoscopies (e.g. due to obstructions or NSAID enteropathy) as determined by physician discretion.

f. Has a cardiac device (e.g. pacemaker or ICD-Implantable Cardioverter Defibrillator) or any other active implanted device g. Known sensitivity to iodine, or with known kidney failure. h. Known condition which precludes compliance or is contraindicated with study and/or device instructions.

i. Has a Magnetic Image Resonance (MRI) procedure scheduled within 1 month j. Known condition of drug abuse and/or alcoholism. k. Women who are either pregnant or nursing at the time of screening (to be verified by urine or serum pregnancy test for woman of child- bearing potential who are not post-menopausal or undergone surgical sterilization.

l. Concurrent participation in another clinical trial using any investigational drug or device.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Gross, Principal Investigator — NYU Langone Health
Locations (1):
- Mayoclinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- C-Scan Procedure: Subjects who are at high or at average risk for developing CRC and who are scheduled for optical colonoscopy will undergo C-Scan procedure
  C-Scan procedure: The subjects will be connected to the C-Scan Track and after successful system's activation. The subject will be asked to ingest the C-Scan Capsule with some water, contrast media The subject will be required to ingest daily dose (3 X 15 ml) of contrast media. Capsule procedure is completed upon capsule excretion.
  o Collecting procedure related data: Technical performance in normal daily routine, Segmental transit time,Procedure duration, Number of Bowel movements , Similarity between C-Scan results and colonoscopy Etc,
Period: Overall Study
Arm/Group | C-Scan Procedure
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: High risk and average risk for CRC
Arm/Group | C-Scan Procedure
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race: American Indian or Alaska Native | 0
  race: Asian | 1
  race: Caucasian | 34
  race: African American | 3
  race: Unknown | 2
  race: More than one race | 0
Belly Circumference [Mean (Standard Deviation); unit: Centimeters] | 95.6 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Incidence of Device and Procedure Related Serious Adverse Events (SAE)
Description: The safety of the Check-Cap System will be evaluated by the incidence of device and procedure related Serious Adverse Events (SAE), as adjudicated by the Independent Physician Adjudicator.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | C-Scan Procedure
Number analyzed (Participants) | 40
Participants | 0

2. Secondary Outcome: Non-compliance Rate of Subjects (%)
Description: Subject compliance will be assessed by
  - Non-compliance rate throughout the study via diary completion by the subject Specific questionnaire. completed by remote subject monitoring (via telephone) The rate will be measured in a percentage scale (1-100%) Score less then 50% will be considered as a compliance failure
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | C-Scan Procedure
Number analyzed (Participants) | 40
Participants | 40

3. Secondary Outcome: To Evaluate Subject's Satisfaction
Description: Subject satisfaction will be established by:
  Designated questionnaire that focuses on patient's impressions regarding tolerance and potential safety concerns, which will be provided to the subjects after the C-Scan procedure and after the colonoscopy procedure. Acceptance criteria was defined as average score >3.5 (1- low satisfaction to 5- high satisfaction), which represent high satisfaction with the safety and tolerance of the C-scan system.
  Comparing patient's satisfaction with C-Scan procedure and colonoscopy procedure
Time Frame: 8 weeks
Population: The C-scan questionnaire was completed following the excretion of the C-Scan capsule. Forty subjects completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-Scan Procedure
Number analyzed (Participants) | 40
units on a scale | 3.42 (1.25)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event were reported to the study nurse and or study PI
Arm/Group | C-Scan Procedure
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 13/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C-Scan Procedure (N=40)
Abdominal pain, cramps (Gastrointestinal disorders) | 8 (8)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3)
diarrhea / soft stool (Gastrointestinal disorders) | 2 (2)
Superficial Phlebitis (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed publications and presentations by the Investigator, the Institution or their personnel and associates, resulting from or relating to the Study, must be submitted to the Company for review and approval at least forty five (45) days prior to submission for publication or presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT03735407/Prot_SAP_000.pdf